CLINICAL TRIAL: NCT05381181
Title: Clinical Study of the Safety and Efficacy of Next-generation Universal CD19 Chimeric Antigen Receptor T Cells in the Treatment of Relapsed or Refractory B Cell Malignancies
Brief Title: Safety and Efficacy Evaluation of Next-generation CD19-UCART
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-BRL-301
Record Dates: First submitted 2022-05-11; First posted 2022-05-19 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-05

CONDITIONS: Acute Lymphoblastic Leukemia; Non Hodgkin Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-UCART (Experimental): All patients will be treated with at least 1 injection of CD19- UCART. A dose of 5x10^6/kg BW of CD19-UCART will be evaluated. If > 1/6 of DLT occurred, the dose would be reduced to 2.0x10^6/kg BW.
  Interventions: Biological: CD19-UCART

INTERVENTIONS:
Biological: CD19-UCART — A conditioning therapy with cyclophosphamide and fludarabine will be conducted before CD19-UCART injection. VP16 can be added to the conditioning therapy.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Next-generation CD19-UCART in patients with relapsed or refractory B-cell hematological malignancies.

DETAILED DESCRIPTION:
CD19-UCART is a kind of "off-the-shelf" product originated from health donor's PBMC. This is an open-label, single arm study to evaluate the safety and anti- tumor efficacy of Next-generation CD19-UCART in the treatment of relapsed or refractory B-cell hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary to participate in this clinical study and sign informed consent form;
2. The expected survival period is at least three months;
3. There is no other severe cardiopulmonary disease, and the liver and kidney function are normal (except for the subject with tumor lesions in the liver and kidney);
4. Patients cannot benefit from autologous CAR-T cell therapy due to T cell separation failure or CART amplification failure in the preparation of autologous CART, or the failure to complete apheresis or disease progression; Or the content of T cells in PBMC of peripheral blood is less than or equal to 10%; Or the disease is not effectively controlled within one month after autologous CAR-T transfusion, and the patient cannot receive CAR-T transfusion again;
5. The test results show that CD19 is positive in the tumor;
6. Patients with relapsed or refractory CD19-positive acute B-lymphocyte leukemia or B-cell non-Hodgkin's lymphoma. Patients with r/r B-ALL: 1 years old ≤ patient age ≤60 years. Patients with r/r B-NHL: 18 years old ≤ patient age ≤65 years old
7. Hematological indicators meet the following conditions: 1) WBC count ≥ 1.5× 10^9/L; 2) Absolute value of neutrophils ≥ 0.8× 10^9/L; 3) Lymphocyte count ≥ 0.1× 10^9/L; 4) Hemoglobin ≥ 60 g/L; 5) Platelet count ≥ 20× 10^9/L;
8. Blood biochemistry shall meet the following requirements 1) or 2): 1) patients with liver and kidney without tumor lesions: A) Total bilirubin (TBIL)≤1.5*ULN (upper limit of normal value), unless suffering from Gilbert's syndrome; B) aspartate aminotransferase (AST) ≤ 1.5 * ULN; C) ALT ≤ 1.5 * ULN; D) Scr ≤ 1.5 * ULN; E) Urea (URA) ≤ 1.5 * ULN; 2) patients with liver and kidney tumor lesions: a) TBIL≤5*ULN； b) AST≤5*ULN； c) ALT≤5*ULN； d) SCr≤5*ULN； e) Urea≤5*ULN；
9. Heart function: good hemodynamic stability, and the left ventricular ejection fraction (LVEF) is higher than or equal to 55%;
10. Serum viruses such as HIV, TP, HBV(HBV-DNA) and HCV(HCV-DNA) are all negative;
11. ECOG activity status score: 0-2 points;
12. Accept the requirement that effective contraception be used throughout the study;
13. Willing to abide by the rules established in this study.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Having a pregnancy plan in the next two years;
3. Has received graft-versus-host disease treatment in the past;
4. Has received allogeneic cell therapy in the past 6 weeks;
5. Has received allogeneic stem cell transplantation within the past 6 months;
6. Individual extramedullary relapse B-ALL;
7. Suffering from severe mental disorder;
8. Active autoimmune diseases requiring immunotherapy;
9. Has suffered from other malignant tumors in the past;
10. Patients with severe cardiovascular disease;
11. Prothrombin time or activated partial thromboplastin time or international normalized ratio > >1.5*ULN； in the absence of anticoagulant therapy;
12. There is active infectious disease or need any major infection events of high-level antibiotics; 13. Any condition that, in the opinion of the investigator, may increase the subject's risk or interfere with the study results.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) incidence | Day 0 up to 35 days after T cell infusion
  Incidence of adverse events (AEs) defined as DLTs

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At 12 weeks
  Proportion of patients in whom a response among complete response and partial response as defined by standard disease-specific criteria, will be observed.

OTHER OUTCOMES:
Duration of response (DOR) | up to 2 years after T cell infusion
  DOR is defined as the time from the first objective response to disease progression or death due to disease relapse or drug-related toxicity
Progress free survival (PFS) | up to 2 years after T cell infusion
  PFS is defined as the time from the T cell infusion date to the date of disease progression or death from any cause
Overall survival (OS) | up to 2 years after T cell infusion
  OS is defined as the time from the date of leukapheresis until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Prof., Principal Investigator — The First Affiliated Hospital of Zhengzhou University

IPD SHARING:
Plan to Share IPD: No